CLINICAL TRIAL: NCT01027741
Title: Integrating Cancer Control Referrals and Navigators Into United Way 211 Missouri
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: United Way Missouri (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 000708
Record Dates: First submitted 2009-12-04; First posted 2009-12-09 (Estimated); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Phone Referral (Experimental): Participants receive phone referral to cancer control and prevention services.
  Interventions: Behavioral: Phone Referral
- Tailored Cancer Communication (Experimental): Participants will receive phone referral to cancer control and prevention services as well as tailored materials in the mail.
  Interventions: Behavioral: Phone Referral; Behavioral: Tailored Cancer Communication
- Cancer Control Navigator (Experimental): Participants will receive phone referral to cancer control and prevention services as well as a personal cancer control navigator.
  Interventions: Behavioral: Phone Referral; Behavioral: Cancer Control Navigator
- Control (No Intervention): Participants receive only recommendation to talk to health care professional.

INTERVENTIONS:
Behavioral: Phone Referral — Participants receive phone referral to cancer control and prevention services.
  Arms: Cancer Control Navigator; Phone Referral; Tailored Cancer Communication
Behavioral: Tailored Cancer Communication — Mailed material with messages tailored to participant's age, gender, race/ethnicity, whether he or she has kids in the home, reason for calling 211, and cancer control need.
  Arms: Tailored Cancer Communication
Behavioral: Cancer Control Navigator — A cancer control navigator is assigned to each participant. This navigator helps the participant make and keep cancer control and prevention appointments, as well as providing resources and guidance to help address participant barriers to use of needed cancer control and prevention services. Intervention is phone-based.
  Arms: Cancer Control Navigator

SUMMARY:
The proposed study will:

1. estimate the prevalence of need for cancer screening and prevention in a population of 211 callers;
2. determine whether cancer communication interventions delivered through 211 can increase use of breast, cervical and colon cancer screening, HPV vaccination, smoking cessation and adoption of smoke free home policies;
3. determine how intensive an intervention is needed to bring about these changes; and
4. determine whether the effectiveness of these interventions is enhanced when callers' basic needs have been addressed. Connecting these systems - 211, clinical and community cancer control programs and navigation services - should benefit disadvantaged Americans. The proposed study will evaluate the effects of this approach to eliminating cancer disparities.

We hypothesize that the proportion of 211 callers who obtain a needed cancer control service will:

1. differ significantly by study group as follows: N > T > P > CONTROL;
2. vary significantly across study groups based on the intervention dose callers receive; and
3. vary significantly across study groups based on whether callers' original need was resolved, the extent of their basic needs, and their perception of life as manageable and predictable (i.e., sense of coherence).

(Dissemination Aim): Determine costs to 211 and effects on quality of service by offering cancer control referrals.

DETAILED DESCRIPTION:
For Americans living in poverty, cancer prevention and screening is a lower priority than meeting basic needs. When basic needs are addressed, the likelihood of engaging in these preventive behaviors increases. Strategies to eliminate cancer disparities in disadvantaged populations must recognize and address this fundamental challenge. We propose the first-ever cancer communication research partnership with United Way 2-1-1, a telephone information and referral system reaching millions of low-income and minority Americans every year and connecting them to locally available resources that can meet their basic needs. By proactively linking these callers to evidence-based cancer control services available for free in their community, cancer disparities could be reduced.

The proposed study will:

1. estimate the prevalence of need for cancer screening and prevention in a population of 211 callers;
2. determine whether cancer communication interventions delivered through 211 can increase use of breast, cervical and colon cancer screening, HPV vaccination, smoking cessation and adoption of smoke free home policies;
3. determine how intensive an intervention is needed to bring about these changes; and
4. determine whether the effectiveness of these interventions is enhanced when callers' basic needs have been addressed. Connecting these systems - 211, clinical and community cancer control programs and navigation services - should benefit disadvantaged Americans. The proposed study will evaluate the effects of this approach to eliminating cancer disparities.

Objectives:

Study group assignment -- By random assignment they will then receive either:

* Tailored Cancer Communication to help them act on the cancer control referral they received;
* A Cancer Control Navigator to help them overcome obstacles to obtaining needed cancer control services;
* Cancer Control Phone Referral Only; or,
* No intervention control

The study aims are to:

1. Estimate the prevalence of need for cancer screening and prevention in a population of 211 callers and compare these rates to population data from Missouri and the U.S.
2. Evaluate effects of Tailored Cancer Communication (T), Cancer Control Navigation (N), Cancer Control Phone Referral Only (P) on use of cancer control services in a randomized trial among 211 callers.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* caller to 211 who was randomly allocated to one of two study-specific information specialists
* resident of Missouri
* calling for unmet needs for self

Exclusion Criteria:

* calling on behalf of client or other person

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4762 (Actual)
Dates: Start 2009-12 (Actual); Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Use of cancer screening and preventive services | 0ne and four months post-intervention

SECONDARY OUTCOMES:
Resolution of a caller's original problem | One month post-intervention
Degree of unmet basic needs | One and four months post-intervention
Sense of coherence | One and four months post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Matthew W Kreuter, PhD, MPH, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University in St. Louis, St Louis, Missouri, United States